CLINICAL TRIAL: NCT00194233
Title: Serum and Peritoneal Fluid Bank for Assessment of Markers of Endometriosis
Brief Title: Serum and Peritoneal Fluid Bank for Endometriosis Markers
Status: Completed | Type: Observational
Sponsor: University of Pennsylvania (Other)
Responsible Party: Kurt T Barnhart, MD, MSCE, University of Pennsylvania
Other Study IDs: 708870; RRU008
Record Dates: First submitted 2005-09-13; First posted 2005-09-19 (Estimated); Last update posted 2016-08-16 (Estimated); Status verified 2016-08

CONDITIONS: Endometriosis
Keywords: Endometriosis
MeSH Terms: conditions — Endometriosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum, Plasma, Peritoneal fluid

SUMMARY:
The purpose of this study is to investigate differences in protein expression profiles of blood and peritoneal fluid samples obtained from patients who do, and those who do not, have endometriosis seen during laparoscopic surgery. These profiles may include both known and novel markers for diagnosing endometriosis.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing laparoscopic surgery for one of the following indications:

  1. infertility
  2. pain
  3. tubal sterilization
* For cases, visualization of endometriosis
* For controls, absence of endometriosis

Exclusion Criteria:

* None

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Women undergoing Laparoscopy at HUP
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2003-11; Primary Completion 2007-01 (Actual); Study Completion 2008-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kurt T Barnhart, MD, MSCE, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania Reproductive Research Unit, Philadelphia, Pennsylvania, United States